CLINICAL TRIAL: NCT07120139
Title: Clinical Effectiveness of Episodic Use of Bioactive Silica Based Versus Continuous Use of Fluoride Desensitizing Toothpastes in Management of Dentin Hypersensitivity (A 6m Randomized Clinical Trial)
Brief Title: Clinical Effectiveness of Episodic Use of Bioactive Silica Based Versus in Management of Dentin Hypersensitivity (A 6m Randomized Clinical Trial)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rawda Hesham Abd ElAziz (Other)
Responsible Party: Sponsor-Investigator, Rawda Hesham Abd ElAziz, Associate Professor, Conservative dentistry department, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CONS2R
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Dentin Hypersensitivity
Keywords: Bioactive Silica Based with calcium booster (Refix technology) toothpaste; Dentin hypersensitivity.
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 Episodic use of Refix booster Bioactive Silica with calcium booster toothpaste (Experimental)
  Interventions: Procedure: episodic use of the desensitizing toothpaste
- Group 2: Episodic use of Regenerador Sentitive: Bioactive Silica Based toothpaste, (Experimental)
  Interventions: Procedure: episodic use of the desensitizing toothpaste
- Group 3: Episodic use of (Sensodyne Rapid action) Fluoride containing desensitizing Toothpaste, (Experimental)
  Interventions: Procedure: episodic use of the desensitizing toothpaste
- Group 4: Continuous use of (Sensodyne Rapid action) Fluoride containing desensitizing Toothpaste (Active Comparator)
  Interventions: Procedure: continuous use of the conventional desensitizing toothpaste

INTERVENTIONS:
Procedure: episodic use of the desensitizing toothpaste — subjects assigned to episodic treatment will use the assigned toothpaste with the same previous instructions for two 8-week treatment periods, followed by an 8-week phase in which they will use the conventional fluoride dentifrice (Signal Complete 8 Original, Unilever, Egypt), which has no documented desensitizing efficacy
  Arms: Group 1 Episodic use of Refix booster Bioactive Silica with calcium booster toothpaste; Group 2: Episodic use of Regenerador Sentitive: Bioactive Silica Based toothpaste,; Group 3: Episodic use of (Sensodyne Rapid action) Fluoride containing desensitizing Toothpaste,
Procedure: continuous use of the conventional desensitizing toothpaste — The patients will be instructed to use 1 inch amount of the assigned desensitizing toothpaste and soft bristle toothbrushes with the same brushing technique they will be taught in the intervention visit for 2 minutes twice a day (morning and last thing at night ) without further rinsing, only spitting of the excess material every day along the whole study period for the continuous treatment group.
  Arms: Group 4: Continuous use of (Sensodyne Rapid action) Fluoride containing desensitizing Toothpaste

SUMMARY:
The aim of the study to compare the clinical effectiveness of Episodic use of Bioactive Silica Based versus continuous use of fluoride based desensitizing toothpastes in management of dentin hypersensitivity (DH) of adult patients over 6m follow up and evaluating patient satisfaction regarding the treatment provided. Episodic use will be tested as it reflects the effectiveness in a clinical scenario regarding patient compliance and adherence to the treatment where some of the Egyptian patients stop the treatment once improvement occurs due to financial constraints

ELIGIBILITY:
Inclusion Criteria:

Patients with DH, VAS ≥ 3 and Schiff sensitivity score needed to be ≥2, indicating that application of a jet of air makes the patient respond and move or requests discontinuation of the stimuli application.

• Teeth with DH related to Non- carious Cervical lesions (abrasion, abfracture, erosion).

• Teeth with gingival recession and exposed root dentin.

-

Exclusion Criteria:

* Patients with known allergies or adverse reactions to any ingredient of the tested materials.

Systematic disease and/ or physical disabilities that may affect participation. • Patients who did any periodontal surgeries within the previous 3 months.

• Patients with orthodontic appliances, or restorative work that might interfere with evaluation.

• Patient who frequently use analgesics or any drugs that could affect the pain level.

• Home or in-office bleaching and/ or in office fluoride application for 6 months before beginning of treatment.

• Pregnant females with frequent vomiting attacks.

• Smokers.

• Systemic conditions that cause or predispose patients to develop dentin hypersensitivity (for example, gastroesophageal reflux disease, GERD).

• Excessive dietary or environmental exposure to acids.

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Degree of Dentin hypersensitivity | change from the baseline, 1month, 2months, 4 months, 6 months after treatment
  Visual analog scale (VAS)

SECONDARY OUTCOMES:
Examiner Assessment to level of patient pain | change from the baseline, 1month, 2months, 4 months, 6 months after treatment
  Schiff sensitivity scale [SSS]
Patient satisfaction with the Treatment | change from the baseline, 1month, 2months, 4 months, 6 months after treatment
  4-point Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No